CLINICAL TRIAL: NCT06178770
Title: Injection Intervals in Real-world Neovascular Age-related Macular Degeneration (nAMD) Patients Switching to Brolucizumab With at Least 12 Months of Follow-up
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRTH258A2018
Record Dates: First submitted 2023-12-12; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: nAMD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (5):
- Overall cohort
- 12-month BRO cohort
- 18-month BRO cohort
- 12-month ALT cohort
- 18-month ALT cohort

SUMMARY:
This retrospective study included nAMD patients whose eyes were grouped into the following cohorts, with the overall cohort receiving ≥ 1 brolucizumab injection; the 12-month and 18-month brolucizumab (BRO) cohorts, which consisted of nAMD patient eyes who switched from a previous anti-vascular endothelial growth factor (VEGF) and had ≥3 brolucizumab injections with no other anti-VEGF in the first 12 months (360 days) and 18 months (540 days) of follow-up respectively; and the 12-month and 18-month alternating (ALT) cohorts, which consisted of nAMD patient eyes who switched from a previous anti-VEGF to brolucizumab and had ≥2 brolucizumab injections and ≥1 injection of another anti-VEGF in the first 12 months and 18 months of follow-up, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of nAMD.
* Patients were on a previous anti-VEGF therapy and then switched to brolucizumab.
* Patients remained on brolucizumab for at least 12 months.
* Patients had exactly 360 days or more of follow-up after first brolucizumab injection.
* For BRO cohort only: Patients received at least three injections of brolucizumab during study period.
* For ALT cohort only: Patients received at least two injections of brolucizumab and one injection of another anti-VEGF during the study period.

Exclusion Criteria:

* For BRO cohort only: Patients who received any other anti-VEGF therapy during the 12-month follow-up period.
* Eyes missing bilaterality information in their nAMD diagnosis.
* Eyes missing bilaterality information in their brolucizumab injections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 414 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Mean change in injection interval from baseline to Month 12 for BRO and ALT cohorts | Baseline, Month 12

SECONDARY OUTCOMES:
Change in injection interval from first brolucizumab injection to Month 18 for BRO and ALT cohorts | Baseline, Month 18
Change in visual acuity (VA) from first brolucizumab injection to Month 12 (for BRO and ALT cohorts) and Month 18 (for BRO cohort) | Baseline, Months 12 and 18
Change in central macular thickness (CMT) from first brolucizumab injection to Month 12 (for BRO and ALT cohorts) and Month 18 (for BRO cohort) | Baseline, Months 12 and 18
Age | Baseline
Gender | Baseline
Visual acuity (Early Treatment Diabetic Retinopathy Study [ETDRS] Letters) | Baseline, Month 12 and Month 18
Anti-VEGF treatment status | Baseline
Last injection interval before switch to brolucizumab in prior-treated eyes | Baseline
Central macular thickness (CMT) | Baseline, Month 12 and Month 18
Intraretinal fluid (IRF) | Baseline
Subretinal fluid (SRF) | Baseline
Pigment epithelial detachment (PED) | Baseline
Number of brolucizumab injections and non-brolucizumab injections from first brolucizumab injection to 12 months (for ALT cohort) | Baseline, Month 12
Ocular adverse events (AEs) in eyes treated with at least one brolucizumab injection | Up to 3 years
Median time (days) from first brolucizumab injection to AE | Up to 3 years
Median time (days) from last brolucizumab injection pre-AE to AE | Up to 3 years
Median time (days) from AE to resolution | Up to 3 years
Median number of brolucizumab injections pre-AE including the index injection | Up to 3 years
Proportion of patients in different levels of vision recovery after AE resolution | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States